CLINICAL TRIAL: NCT02361125
Title: Patient Controlled Administration of Methylphenidate for Cancer Related Fatigue
Brief Title: Patient Controlled Administration of Methylphenidate for Cancer Related Fatigue - PRN Methylphenidate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-166; NCI-2015-00623 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Fatigue
Keywords: Fatigue; Cancer related fatigue; Methylphenidate; Methylphenidate Hydrochloride; Ritalin; Concerta; Fatigue evaluations
MeSH Terms: conditions — Fatigue | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Methylphenidate (Experimental): Participants given a 7 day supply of 5 mg methylphenidate tablets (to take a maximum of 20 mg/day, for total of 28 tablets). Directions for use are to take one 5 mg tablet by mouth as needed every 2 hours for participant described significant fatigue (maximum of 4 tablets/day).
  Evaluation of fatigue, ability to sleep, and general symptom questions at baseline visit, daily while on study drug, and on seventh day of treatment.
  Interventions: Drug: Methylphenidate; Behavioral: Fatigue Evaluations

INTERVENTIONS:
Drug: Methylphenidate — 5 mg tablet by mouth as needed every 2 hours for participant described significant fatigue. Participants to take a maximum of 20 mg/day, for total of 28 tablets for 7 days.
  Other Names: Methylphenidate Hydrochloride; Ritalin; Concerta
Behavioral: Fatigue Evaluations — Participants to have evaluation of their fatigue, ability to sleep, and will answer a set of general symptom questions at baseline visit, daily while on study drug, and on seventh day of treatment.

SUMMARY:
The goal of this clinical research study is to evaluate the effectiveness of ritalin (methylphenidate) taken on an as needed basis for the management of cancer related fatigue. The effects of methylphenidate on pain, mood, and sedation will be evaluated. Researchers will also evaluate the level of fatigue throughout the day and any possible causes of fatigue.

DETAILED DESCRIPTION:
Fatigue is a major problem in cancer patients. Methylphenidate is a drug currently FDA approved for the treatment of attention deficit disorder and narcolepsy (sleep disorder). Methylphenidate has shown a benefit in improving thinking and decreasing drowsiness and pain in cancer patients taking opioids (pain killers). Methylphenidate has also shown a rapid response in treating depression.

Participants in this study will at first have an evaluation of their fatigue, ability to sleep, and they will answer a set of general symptom questions. It will take about 20 minutes to complete the evaluation. Participants will have a blood test called TSH (thyroid-stimulating hormone) performed to rule out the possibility of thyroid dysfunction as cause of fatigue.

The study will last for 7 days. Participants will be able to take up to four methylphenidate tablets a day on an as needed basis for fatigue. Participants will keep a daily diary where they will record their fatigue rating (0-10) before and 2 hours after taking methylphenidate. The research nurse will contact participants daily by phone (in person for in-patients) to make sure the daily diary is being filled out, to ask about side effects of treatment, and to ask participants to rate their fatigue at four times during the past day and about any possible causes of fatigue.

On the 7th day of treatment, participants will be evaluated in the palliative care clinic or by telephone. Evaluation of fatigue, ability to sleep, and general symptoms along with an evaluation of side effects and effectiveness of methylphenidate will be performed. The evaluation will take about 15 minutes to complete. If participants develop intolerable side effects while on study, the medication will be stopped and they will be removed from the study.

If participants find the drug beneficial and wish to continue taking it, they will be given a prescription for methylphenidate and can be followed as an outpatient in the palliative care clinic. Participants who choose to continue the medication will be evaluated at the end of 4 weeks for fatigue, ability to sleep, and general symptoms along with an evaluation of side effects and effectiveness by phone or in the clinic. The evaluation will take about 15 minutes to complete.

This is an investigational study. The use methylphenidate is investigational. A total of 36 patients will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients seen in the outpatient palliative care clinic or inpatients seen by the palliative care consult team or the fatigue clinic.
2. Presence of fatigue on a numerical scale during the last 24 hours of more or equal to 4 on a 0 to 10 scale on which 0 equals no fatigue and 10 worst possible fatigue.
3. Patient should describe fatigue as being present for a minimum of four days.
4. If patients are on opioids for the treatment of cancer pain, they must have had no dose changes (>25%) for at least 48 hours prior to study entry. Change in opioid dose after study entry is allowed.
5. Presence of relatively intact cognition defined by normal Mini Mental State Questionnaire according to age and education level. A score of 24 or above is usually considered normal.
6. Signed written informed consent.
7. Patient must be 18 years or older.The questionnaires used in this study have been validated only in the adult population.
8. Patient willing to keep a daily fatigue diary, engage in daily telephone follow up with a nurse and after 7 days of treatment either return for a follow up visit or this can be done over the telephone.
9. Hemoglobin of >/=10 g/dl within 2 weeks of enrollment. If the patient has not had blood drawn for a hemoglobin level in the past two weeks, one will be done to determine the eligibility.

Exclusion Criteria:

1. Major contraindication to methylphenidate i.e. hypersensitivity
2. Currently on methylphenidate or has been on methylphenidate within the last 10 days.
3. Inability to complete the baseline assessment forms or to understand the recommendations for participation in the study.
4. Pregnant or lactating women. Childbearing age women are not on birth control.
5. Patients taking MAO inhibitors, tricyclic antidepressants, clonidine, psychostimulants, concurrent steroids or other medications specifically for fatigue
6. Patients with glaucoma, history of marked anxiety disorder, or history of substance abuse.
7. CAGE questionnaire score is 2 or above on a 0 to 4 scale.
8. Patients with history of seizures or uncontrolled CNS disease, significant hepatic or renal dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2002-08-01 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Fatigue Measurement on a 10-point scale | 7 days
  Primary endpoint is fatigue as measured on a 10-point scale. An average 2-point reduction in fatigue from before to 2 hours after taking methylphenidate considered a clinical success.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org